CLINICAL TRIAL: NCT02983214
Title: Study of the Efficacy and Safety of Cilostazol in the Prevention of Ischemic Vascular Events in Diabetic Patients With Symptomatic Peripheral Artery Disease.
Brief Title: Diabetic Artery Obstruction: is it Possible to Reduce Ischemic Events With Cilostazol?
Acronym: DORIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ioannina (Other)
Collaborators: LIBYTEC Pharmaceutical S.A. (Unknown)
Responsible Party: Principal Investigator, Alexandros Tselepis, Professor of Biochemistry and Clinical Chemistry, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Cilo-UoI-2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Ischemic Stroke; Peripheral Artery Disease; Diabetes Mellitus, Type 2
Keywords: Cilostazol; Clopidogrel; Peripheral Artery Disease
MeSH Terms: conditions — Ischemic Stroke; Peripheral Arterial Disease; Diabetes Mellitus, Type 2 | interventions — Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator): Clopidogrel 75 mg/day
  Interventions: Drug: Clopidogrel
- Clopidogrel plus cilostazol (Active Comparator): Clopidogrel 75 mg/day plus cilostazol 100 mg twice/day
  Interventions: Drug: Clopidogrel; Drug: Cilostazol

INTERVENTIONS:
Drug: Clopidogrel
  Other Names: Plavix, Clodelib, Clovelen
Drug: Cilostazol
  Other Names: Claudiasil
  Arms: Clopidogrel plus cilostazol

SUMMARY:
Investigation of the clinical efficacy and safety of dual antiplatelet therapy with clopidogrel and cilostazol versus clopidogrel alone in preventing ischemic vascular events in patients with type 2 diabetes and symptomatic peripheral arterial disease.

DETAILED DESCRIPTION:
Cilostazol is a quinoline derivative that selectively and reversibly inhibits cellular cyclic adenosine monophosphate (cAMP) phosphodiesterase III, thus suppressing cAMP degradation and maintaining its high intracellular levels. Through this mechanism, cilostazol inhibits platelet aggregation, exerting significant antiplatelet and antithrombotic activity. Cilostazol also improves endothelial function and exerts anti-inflammatory, anti-atherogenic and vasodilatory effects. Additionally, cilostazol inhibits equilibrative nucleoside transporter-1 (ENT-1) which is responsible for the cellular uptake of adenosine, reducing its plasma concentration. Through this mechanism, cilostazol maintains high extracellular adenosine concentration allowing adenosine to exert its biological effects. Thus, cilostazol not only shows potent antithrombotic activity, but also prevents restenosis after percutaneous coronary intervention (PCI). Finally, cilostazol has beneficial effects in the lipidemic profile reducing triglyceride levels and increasing HDL-cholesterol. Clinical studies have shown that in patients with intermittent claudication, cilostazol increases the walking distance. Based on these studies, cilostazol administration in combination with an antiplatelet drug (clopidogrel or aspirin) is recommended for patients with intertermittent claudication.

Recent pharmacodynamic studies have demonstrated that adding cilostazol to aspirin or clopidogrel may represent an effective way to overcome high on-treatment platelet reactivity. Additionally, clinical studies have shown that the addition of cilostazol to dual antiplatelet therapy with aspirin and clopidogrel (triple antiplatelet therapy, TAPT) in patients with acute coronary syndrome undergoing PCI offers significant clinical benefit. This favorable effect of cilostazol was confirmed in a recent meta-analysis which included nine studies and a total of 2,179 patients undergoing PCI. Furthermore, other clinical studies have shown that administration of TAPT with cilostazol reduces restenosis after PCI. Finally, the administration of dual antiplatelet therapy with cilostazol and aspirin significantly reduces the progression of symptomatic intracranial arterial stenosis compared to monotherapy with aspirin.

The aim of The Diabetic artery Obstruction: is it possible to Reduce Ischemic events with Cilostazol? (DORIC) trial is to investigate the clinical efficacy and safety of dual antiplatelet therapy (DAPT) with clopidogrel and cilostazol versus clopidogrel alone in preventing ischemic vascular eventsin patients with type 2 diabetes (DM2) and symptomatic peripheral arterial disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥50 years with DM2 and symptomatic PAD diagnosed clinically (according to Fontaine criteria, stage IIa or IIb and III) and by measuring the ΑΒΙ.

Exclusion Criteria:

* Congestive heart failure, history of ventricular tachycardia, ventricular fibrillation or multifocal ventricular extrasystoles or QTc prolongation.
* Patients with atrial fibrillation taking any anticoagulant therapy or patients with a history of cardioembolic ischemic stroke or hemorrhagic stroke.
* Patients with a history (≤ 12 months) of acute coronary syndrome receiving dual antiplatelet therapy, or patients receiving monotherapy with aspirin.
* Patients with hepatic impairment (child-Pugh staging, calibration ≥ 5) or renal impairment (creatinine clearance ≤ 30ml / min), recent peptic ulcer, a history of hypersensitivity to cilostazol, cancer patients undergoing treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who suffer from the primary efficacy end point which is composite of acute ischemic stroke/transient ischemic attack (TIA), myocardial infarction (MI), or death from vascular causes during the entire follow-up period. | 12 months
  Death from vascular causes: cardiovascular or cerebrovascular
Number of participants who suffer from bleeding events as defined by the Bleeding Academic Research Consortium (BARC) criteria during the entire follow-up period. | 12 months

SECONDARY OUTCOMES:
Number of participants whose major secondary efficacy end point desribed in the description section is observed. | 12 months
  Acute ischemic stroke / TIA, AMI, coronary stent thrombosis, PCI, coronary restenosis, death from cardiovascular causes, death from any cause, hospitalization for acute limb ischemia, lower extremity arterial revascularization, improvement of ABI and pain-free walking distance values.
Number of participants who suffer from the secondary safety end points which are palpitations, tachycardia, headache, diarrhea, urticaria, neoplasms, blood disorders, drug interruption. | 12 months
  Blood disorders: transient thrombocytopenia, leukopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Atherothrombosis Research Centre / Laboratory of Biochemistry, University of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalantzi KI, Tsoumani ME, Goudevenos IA, Tselepis AD. Pharmacodynamic properties of antiplatelet agents: current knowledge and future perspectives. Expert Rev Clin Pharmacol. 2012 May;5(3):319-36. doi: 10.1586/ecp.12.19. PMID 22697594
- [Background] Dindyal S, Kyriakides C. A review of cilostazol, a phosphodiesterase inhibitor, and its role in preventing both coronary and peripheral arterial restenosis following endovascular therapy. Recent Pat Cardiovasc Drug Discov. 2009 Jan;4(1):6-14. doi: 10.2174/157489009787260025. PMID 19149700
- [Background] Jeong YH, Tantry US, Bliden KP, Gurbel PA. Cilostazol to overcome high on-treatment platelet reactivity in korean patients treated with clopidogrel and calcium-channel blocker. Circ J. 2011;75(11):2534-6. doi: 10.1253/circj.cj-11-1076. Epub 2011 Oct 5. No abstract available. PMID 21970840
- [Background] Rizzo M, Corrado E, Patti AM, Rini GB, Mikhailidis DP. Cilostazol and atherogenic dyslipidemia: a clinically relevant effect? Expert Opin Pharmacother. 2011 Mar;12(4):647-55. doi: 10.1517/14656566.2011.557359. Epub 2011 Feb 2. PMID 21284580
- [Background] Liu Y, Fong M, Cone J, Wang S, Yoshitake M, Kambayashi J. Inhibition of adenosine uptake and augmentation of ischemia-induced increase of interstitial adenosine by cilostazol, an agent to treat intermittent claudication. J Cardiovasc Pharmacol. 2000 Sep;36(3):351-60. doi: 10.1097/00005344-200009000-00011. PMID 10975593
- [Background] Tselepis AD. Cilostazol-based triple antiplatelet therapy in the era of generic clopidogrel and new potent antiplatelet agents. Curr Med Res Opin. 2014 Jan;30(1):51-4. doi: 10.1185/03007995.2013.850070. Epub 2013 Oct 18. No abstract available. PMID 24089998
- [Background] Chapman TM, Goa KL. Cilostazol: a review of its use in intermittent claudication. Am J Cardiovasc Drugs. 2003;3(2):117-38. doi: 10.2165/00129784-200303020-00006. PMID 14727939
- [Background] Rooke TW, Hirsch AT, Misra S, Sidawy AN, Beckman JA, Findeiss LK, Golzarian J, Gornik HL, Halperin JL, Jaff MR, Moneta GL, Olin JW, Stanley JC, White CJ, White JV, Zierler RE; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology; Society for Vascular Medicine; Society for Vascular Surgery. 2011 ACCF/AHA Focused Update of the Guideline for the Management of Patients With Peripheral Artery Disease (updating the 2005 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2011 Nov 1;58(19):2020-45. doi: 10.1016/j.jacc.2011.08.023. Epub 2011 Oct 6. No abstract available. PMID 21963765
- [Background] Spiliopoulos S. Antiplatelet therapy in critical limb ischemia: update on clopidogrel and cilostazol. J Cardiovasc Surg (Torino). 2014 Oct;55(5):631-40. Epub 2014 May 28. PMID 24866775
- [Background] Chen Y, Zhang Y, Tang Y, Huang X, Xie Y. Long-term clinical efficacy and safety of adding cilostazol to dual antiplatelet therapy for patients undergoing PCI: a meta-analysis of randomized trials with adjusted indirect comparisons. Curr Med Res Opin. 2014 Jan;30(1):37-49. doi: 10.1185/03007995.2013.850067. Epub 2013 Oct 18. PMID 24083626
- [Background] Min PK, Jung JH, Ko YG, Choi D, Jang Y, Shim WH. Effect of cilostazol on in-stent neointimal hyperplasia after coronary artery stenting: a quantative coronary angiography and volumetric intravascular ultrasound study. Circ J. 2007 Nov;71(11):1685-90. doi: 10.1253/circj.71.1685. PMID 17965485
- [Background] Douglas JS Jr, Holmes DR Jr, Kereiakes DJ, Grines CL, Block E, Ghazzal ZM, Morris DC, Liberman H, Parker K, Jurkovitz C, Murrah N, Foster J, Hyde P, Mancini GB, Weintraub WS; Cilostazol for Restenosis Trial (CREST) Investigators. Coronary stent restenosis in patients treated with cilostazol. Circulation. 2005 Nov 1;112(18):2826-32. doi: 10.1161/CIRCULATIONAHA.104.530097. Epub 2005 Oct 24. PMID 16246948
- [Background] Kwon SU, Cho YJ, Koo JS, Bae HJ, Lee YS, Hong KS, Lee JH, Kim JS. Cilostazol prevents the progression of the symptomatic intracranial arterial stenosis: the multicenter double-blind placebo-controlled trial of cilostazol in symptomatic intracranial arterial stenosis. Stroke. 2005 Apr;36(4):782-6. doi: 10.1161/01.STR.0000157667.06542.b7. Epub 2005 Mar 3. PMID 15746463
- [Background] Panagiotakos DB, Georgousopoulou EN, Pitsavos C, Chrysohoou C, Metaxa V, Georgiopoulos GA, Kalogeropoulou K, Tousoulis D, Stefanadis C; ATTICA Study group. Ten-year (2002-2012) cardiovascular disease incidence and all-cause mortality, in urban Greek population: the ATTICA Study. Int J Cardiol. 2015 Feb 1;180:178-84. doi: 10.1016/j.ijcard.2014.11.206. Epub 2014 Nov 26. PMID 25463360
- [Background] Toyoda K, Uchiyama S, Hoshino H, Kimura K, Origasa H, Naritomi H, Minematsu K, Yamaguchi T; CSPS.com Study Investigators. Protocol for Cilostazol Stroke Prevention Study for Antiplatelet Combination (CSPS.com): a randomized, open-label, parallel-group trial. Int J Stroke. 2015 Feb;10(2):253-8. doi: 10.1111/ijs.12420. Epub 2014 Dec 8. PMID 25487817
- [Derived] Kalantzi K, Tentolouris N, Melidonis AJ, Papadaki S, Peroulis M, Amantos KA, Andreopoulos G, Bellos GI, Boutel D, Bristianou M, Chrisis D, Dimitsikoglou NA, Doupis J, Georgopoulou C, Gkintikas SA, Iraklianou S, Kanellas Kappa, Kotsa K, Koufakis T, Kouroglou M, Koutsovasilis AG, Lanaras L, Liouri E, Lixouriotis C, Lykoudi A, Mandalaki E, Papageorgiou E, Papanas N, Rigas S, Stamatelatou MI, Triantafyllidis I, Trikkalinou A, Tsouka AN, Zacharopoulou O, Zoupas C, Tsolakis I, Tselepis AD. Efficacy and Safety of Adjunctive Cilostazol to Clopidogrel-Treated Diabetic Patients With Symptomatic Lower Extremity Artery Disease in the Prevention of Ischemic Vascular Events. J Am Heart Assoc. 2021 Jan 5;10(1):e018184. doi: 10.1161/JAHA.120.018184. Epub 2020 Dec 17. PMID 33327737